CLINICAL TRIAL: NCT06931678
Title: Evaluation of the Effectiveness of Root Canal Treatment Performed Using Photodynamic Therapy in Teeth With Apical Periodontitis in Patients With Type 2 Diabetes Through Next-Generation Sequencing Microbiome Analysis
Brief Title: Photodynamic Therapy in Root Canal Treatment of T2DM Patients: Microbiome Analysis Via Next-Gen Sequencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKORUCU2; 37379 (Other Grant/Funding Number: Health Institutes of Turkey)
Record Dates: First submitted 2025-04-08; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Necrotic Pulp; Apical Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dental Pulp Necrosis; Periapical Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Necrotic pulped, mature teeth with apical periodontitis (Experimental): This study arm involves the application of antimicrobial photodynamic therapy (aPDT) as an adjunct to conventional root canal treatment in mature permanent teeth diagnosed with apical periodontitis and pulp necrosis. Following standard chemomechanical preparation, methylene blue is used as the photosensitizer, activated by a specific wavelength light source to enhance disinfection of the root canal system.
  Interventions: Procedure: aPDT

INTERVENTIONS:
Procedure: aPDT — This intervention involves the application of antimicrobial photodynamic therapy (aPDT) using methylene blue as a photosensitizer, followed by activation with a light source at an appropriate wavelength. The protocol is applied after conventional root canal preparation and irrigation. The aPDT protocol is standardized and performed in both medically healthy patients and patients with Type 2 Diabetes Mellitus (T2DM), allowing comparison of microbiological and clinical outcomes between the two groups. This intervention aims to enhance root canal disinfection, particularly in anatomically complex areas that are difficult to reach with traditional methods.

SUMMARY:
This clinical study investigates the effectiveness of antimicrobial photodynamic therapy (aPDT) as an additional disinfection method in root canal treatment of patients with Type 2 Diabetes Mellitus (T2DM) who have apical periodontitis (AP). T2DM is known to negatively impact the healing of periapical tissues due to impaired immune response. In this study, methylene blue is used as a photosensitizer, activated by a specific wavelength of light to eliminate residual bacteria that are difficult to reach with conventional cleaning methods. The bacterial load and changes in the root canal microbiome will be analyzed using next-generation sequencing (NGS) of the 16S rRNA gene. The goal is to assess the microbial elimination and healing of periapical lesions, and to improve treatment outcomes in diabetic patients.

DETAILED DESCRIPTION:
Systemic diseases such as Type 2 Diabetes Mellitus (T2DM) are known to influence both the etiology and healing process of endodontic diseases. T2DM is characterized by chronic hyperglycemia and impaired immune responses, which may negatively affect the resolution of periapical inflammation following root canal treatment. Apical periodontitis (AP) is a common endodontic pathology, often resulting from bacterial infection in the root canal system. The prevalence and severity of AP are higher in diabetic patients, and studies have shown reduced survival rates of endodontically treated teeth in this population.

The primary aim of this study is to evaluate the effectiveness of antimicrobial photodynamic therapy (aPDT) as an adjunctive disinfection method following conventional root canal preparation in T2DM patients with AP. aPDT utilizes a photosensitizer-methylene blue in this study-that, when activated by light of a specific wavelength, generates reactive oxygen species to eliminate residual microorganisms in complex anatomical areas such as isthmuses and lateral canals.

The study will utilize next-generation sequencing (NGS) of the 16S rRNA gene to assess bacterial diversity and quantify microbial elimination before and after aPDT application. The healing response of periapical lesions will also be monitored. The findings aim to contribute to improved treatment strategies and outcomes for endodontic therapy in systemically compromised patients, particularly those with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* • Individuals aged between 18 and 65 years

  * Voluntarily agree to participate in the study and attend follow-up sessions
  * Systemically healthy individuals (no systemic diseases)
  * Not taking antihypertensive or antidiabetic medications
  * Not pregnant
  * No use of corticosteroids or antibiotics within the last 3 months
  * No history of smoking
  * No acute pain or extraoral swelling
  * No sinus tract or acute apical abscess
  * Presence of a periapical lesion with a Periapical Index (PAI) score ≥ 3
  * Presence of a mature, single-rooted permanent tooth with completed root development

Exclusion Criteria:

* • Severe periodontal disease

  * Internal or external root resorption
  * Open apex (immature root development)
  * Suspected vertical root fracture
  * Non-restorable teeth
  * Teeth with previous root canal treatment
  * Presence of developmental dental anomalies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
1. Radiographic Assessment of Lesion Healing at 6 months | Postoperative an avarage of 6 months
  Lesion healing will be evaluated using periapical radiographs with the parallel technique, and the Periapical Index (PAI) will be used for the assessment of lesion healing.
Change in Pain Level at day 1, day 3, and day 7 Post-Treatment | Post-Treatment at day 1, day 3, and day 7
  Pain levels will be assessed using the Numerical Rating Scale (NRS), ranging from 0 (no pain) to 100 (worst pain), measured at day 1, day 3, and day 7 post-procedure.

OTHER OUTCOMES:
Microbiome analysis | Posttreatment an average on 3 months
  To assess the impact of aPDT on the root canal microbiota, microbiome analysis will be performed using next-generation sequencing (NGS) of the 16S rRNA gene from samples collected before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hulde Korucu, DDS, Principal Investigator — University of Health Sciences Gülhane Faculty of Dentistry Department of Endodontics
Locations (1):
- Gulhane Faculty of Dentistry, University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The impact of gender differences on pain assessment in the study was also evaluated. Additionally, the effect of age on lesion healing was analyzed. Since the study examines the effects of demographic data on lesion healing and post-treatment pain, demographic data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available for 2 years following the treatment outcomes.